CLINICAL TRIAL: NCT05076604
Title: Effects of Microplegia on Transfusion Rates After Cardiac Surgery: A Randomized Prospective Analysis
Brief Title: Effects of Microplegia on Transfusion Rates After Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Quest Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 201801103
Record Dates: First submitted 2021-10-04; First posted 2021-10-13 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Aortic Valve Disease; Mitral Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Cardioplegic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cardioplegia (Active Comparator): 4:1 cardioplegia consists of 4 parts crystalloid intravenous fluid to one part human blood.
  Interventions: Drug: Cardioplegia Solution
- Microplegia (Active Comparator): Nondiluted microplegia consists of all parts human blood.
  Interventions: Drug: Microplegic Solution No. 1

INTERVENTIONS:
Drug: Cardioplegia Solution — The microplegia solution that is standard of care for all cardiac surgery patients, and which all study subjects will receive is:
  Induction 240 mL Baxter Cardioplegia Solution 10. 5 mL Potassium Chloride 2 meq/ml (21 meq) 250.5 mL total volume
  Maintenance 747 mL Baxter Cardioplegia Solution 3.4 mL Potassium Chloride 2 meq/ml (6.75 meq) 750.4 mL total volume
  Subjects will be randomly assigned to 4:1 cardioplegia or nondiluted microplegia.
  4:1 cardioplegia consists of 4 parts crystalloid intravenous fluid to one part human blood.
  Nondiluted microplegia consists of all parts human blood.
  Arms: Cardioplegia
Drug: Microplegic Solution No. 1 — The microplegia solution that is standard of care for all cardiac surgery patients, and which all study subjects will receive is:
  Induction 240 mL Baxter Cardioplegia Solution 10. 5 mL Potassium Chloride 2 meq/ml (21 meq) 250.5 mL total volume
  Maintenance 747 mL Baxter Cardioplegia Solution 3.4 mL Potassium Chloride 2 meq/ml (6.75 meq) 750.4 mL total volume
  Subjects will be randomly assigned to 4:1 cardioplegia or nondiluted microplegia.
  4:1 cardioplegia consists of 4 parts crystalloid intravenous fluid to one part human blood.
  Nondiluted microplegia consists of all parts human blood.
  Arms: Microplegia

SUMMARY:
This is a prospective, randomized study that is studying the rate of red blood cell (RBC) transfusion rates after planned heart (cardiac) surgery. The study will be conducted at Barnes-Jewish Hospital.

Cardioplegia refers to the method of stopping (arresting) the heart in order to perform heart surgery. However, cardioplegia has also come to refer to the solution to achieve cardiac arrest as well as the machinery in which to deliver the solution. This study will investigate our current Standard Cardioplegia (diluted 4:1 blood cardioplegia) versus Microplegia (undiluted blood cardioplegia) to determine if Microplegia reduces peri-operative blood transfusion rates as compared to Standard Cardioplegia. All forms of cardioplegia will be delivered using the MPS2 Microplegia delivery machine by Quest Medical, Inc.

Patients will be randomized to receive undiluted microplegia or standard 4:1 cardioplegia. The patient and the surgeon will be blinded to the randomization.

Patients will be followed for 30 days post-operatively (or until their initial standard of care post-operative follow up visit with cardiac surgery if that appointment falls outside of the 30 day post-operative window) for the development of any adverse events as well as documentation of blood products given.

We will draw one tube of blood for troponin levels at four time points; 1 draw before surgery (this may be done during the intraoperative period), and 3 draws post-operatively: ICU arrival, 12 hours post-ICU arrival and 24 hours post-ICU arrival. This is to closely monitor the patient for any heart tissue injury.

DETAILED DESCRIPTION:
Cardioplegia was first introduced as a method to protect the heart during cardiac surgery in the 1950s (1). Initially, it consisted of a crystalloid solution and in the 1970s Follette and colleagues proposed that blood was the best mode of delivery of cardioplegia as it is rich in nutrients and oxygen (2). Blood has better osmotic, buffering, and antioxidant qualities that are needed by ischemic myocardium. More recent studies comparing blood and crystalloid cardioplegias showed that there was less cardiac edema, and recovery of ventricular function was more rapid with blood based cardioplegia (3). A meta-analysis of over 5000 patients corroborated these findings and showed that blood based cardioplegia reduced the incidence of postoperative low cardiac output syndrome and was associated with less myocardial damage (4).

Standard diluted blood cardioplegia can also be modified to undiluted blood cardioplegia also known as microplegia. To compare the cardioprotection of 4:1 blood:crystalloid cardioplegia to microplegia, McCann et al randomized 20 pigs to either group. Cardiac edema was measured using histologic morphometrics and echocardiogram. It was noted that both edema percentage and left ventricular mass were significantly more decreased in the microplegia group. Furthermore, all animals receiving microplegia were successfully weaned off cardiopulmonary bypass, whereas only 40% of those receiving standard cardioplegia were successfully weaned (5).

More recently, Algarni et al. showed decreased prevalence of low cardiac output syndrome in patients who received microplegia (n=2,630) (6). Another study compared microplegia and standard cardioplegia in patients undergoing coronary artery bypass grafting and found that the microplegia group had lower troponin levels during the post-operative course. Moreover, microplegia resulted in lower transfusion rates and decreased length of hospital stay (7).

A high rate of patients undergoing cardiac surgery require red blood cell transfusions (RBC). Red blood cell transfusions are strongly associated with both infection and ischemic postoperative morbidity, length of stay, increased early and late mortality, and overall hospital costs (8). Given that previous studies have shown that microplegia is associated with less transfusions, it would be reasonable to incorporate this into practice at Washington University.

ELIGIBILITY:
Inclusion Criteria:

* Are to undergo non-emergent cardiac surgery
* >18 years of age
* Willing and able to provide informed consent

Exclusion Criteria:

* History of endocarditis
* Dialysis-dependent renal failure
* Currently on pre-operative mechanical circulatory support (i.e. ECMO, LVAD or intra-aortic balloon pump [IABP])
* Contraindication to receiving a blood transfusion (i.e. Jehovah's Witness)
* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spencer J Melby, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Follette DM, Fey K, Buckberg GD, Helly JJ Jr, Steed DL, Foglia RP, Maloney JV Jr. Reducing postischemic damage by temporary modification of reperfusate calcium, potassium, pH, and osmolarity. J Thorac Cardiovasc Surg. 1981 Aug;82(2):221-38. PMID 7253686
- [Background] Fremes SE, Christakis GT, Weisel RD, Mickle DA, Madonik MM, Ivanov J, Harding R, Seawright SJ, Houle S, McLaughlin PR, et al. A clinical trial of blood and crystalloid cardioplegia. J Thorac Cardiovasc Surg. 1984 Nov;88(5 Pt 1):726-41. PMID 6387286
- [Background] Guru V, Omura J, Alghamdi AA, Weisel R, Fremes SE. Is blood superior to crystalloid cardioplegia? A meta-analysis of randomized clinical trials. Circulation. 2006 Jul 4;114(1 Suppl):I331-8. doi: 10.1161/CIRCULATIONAHA.105.001644. PMID 16820596
- [Background] McCann UG 2nd, Lutz CJ, Picone AL, Searles B, Gatto LA, Dilip KA, Nieman GF. Whole blood cardioplegia (minicardioplegia) reduces myocardial edema after ischemic injury and cardiopulmonary bypass. J Extra Corpor Technol. 2006 Mar;38(1):14-21. PMID 16637518
- [Background] Algarni KD, Weisel RD, Caldarone CA, Maganti M, Tsang K, Yau TM. Microplegia during coronary artery bypass grafting was associated with less low cardiac output syndrome: a propensity-matched comparison. Ann Thorac Surg. 2013 May;95(5):1532-8. doi: 10.1016/j.athoracsur.2012.09.056. PMID 23608252
- [Background] Onorati F, Santini F, Dandale R, Ucci G, Pechlivanidis K, Menon T, Chiominto B, Mazzucco A, Faggian G. "Polarizing" microplegia improves cardiac cycle efficiency after CABG for unstable angina. Int J Cardiol. 2013 Sep 10;167(6):2739-46. doi: 10.1016/j.ijcard.2012.06.099. Epub 2012 Jul 12. PMID 22795715
- [Background] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460
- [Result] BIGELOW WG, LINDSAY WK, GREENWOOD WF. Hypothermia; its possible role in cardiac surgery: an investigation of factors governing survival in dogs at low body temperatures. Ann Surg. 1950 Nov;132(5):849-66. doi: 10.1097/00000658-195011000-00001. No abstract available. PMID 14771796

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a tertiary care academic medical center.
Pre-assignment Details: All enrolled patients were randomized.
Groups:
- Cardioplegia: 4:1 cardioplegia consists of 4 parts crystalloid intravenous fluid to one part human blood.
  Cardioplegia Solution: The microplegia solution that is standard of care for all cardiac surgery patients, and which all study subjects will receive is:
  Induction 240 mL Baxter Cardioplegia Solution 10. 5 mL Potassium Chloride 2 meq/ml (21 meq) 250.5 mL total volume
  Maintenance 747 mL Baxter Cardioplegia Solution 3.4 mL Potassium Chloride 2 meq/ml (6.75 meq) 750.4 mL total volume
  Subjects will be randomly assigned to 4:1 cardioplegia or nondiluted microplegia.
  4:1 cardioplegia consists of 4 parts crystalloid intravenous fluid to one part human blood.
  Nondiluted microplegia consists of all parts human blood.
- Microplegia: Nondiluted microplegia consists of all parts human blood.
  Microplegic Solution No. 1: The microplegia solution that is standard of care for all cardiac surgery patients, and which all study subjects will receive is:
  Induction 240 mL Baxter Cardioplegia Solution 10. 5 mL Potassium Chloride 2 meq/ml (21 meq) 250.5 mL total volume
  Maintenance 747 mL Baxter Cardioplegia Solution 3.4 mL Potassium Chloride 2 meq/ml (6.75 meq) 750.4 mL total volume
  Subjects will be randomly assigned to 4:1 cardioplegia or nondiluted microplegia.
  4:1 cardioplegia consists of 4 parts crystalloid intravenous fluid to one part human blood.
  Nondiluted microplegia consists of all parts human blood.
Period: Overall Study
Arm/Group | Cardioplegia | Microplegia
Started | 157 | 157
Completed | 136 | 126
Not Completed | 21 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cardioplegia | Microplegia | Total
Number analyzed (Participants) | 157 | 157 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (12.2) | 60.4 (13.4) | 60.7 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 68 | 128
  Male | 97 | 89 | 186
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 17 | 20
  White | 148 | 139 | 287
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 157 | 157 | 314

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative and Postoperative Transfusions
Description: To determine if use of microplegia results in less peri-operative transfusions compared to diluted 4:1 cardioplegia.
Time Frame: Intraoperative (time in operating room), Postoperative (from transfer from operating room to intensive care unit to 30 days)
Measure: Mean (Standard Deviation); unit: units of blood per participant
Arm/Group | Cardioplegia | Microplegia
Number analyzed (Participants) | 157 | 157
units of blood per participant
  Intraoperative Red Blood Cell Transfusion (units) | 2.43 (3.14) | 2.97 (3.49)
  Postoperative Red Blood Cell Transfusion (units) | 4.42 (6.06) | 3.50 (4.25)
Statistical Analysis 1: Comparison: Cardioplegia vs Microplegia; Intraoperative packed red blood cell transfusion; Test type: Superiority; p = 0.354, t-test, 2 sided
Statistical Analysis 2: Comparison: Cardioplegia vs Microplegia; Postoperative red blood cell transfusion; Test type: Superiority; p = 0.314, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cardioplegia | Microplegia
All-Cause Mortality (participants affected / at risk) | 11/157 | 7/157
Serious Adverse Events (participants affected / at risk) | 23/157 | 19/157
Other Adverse Events (participants affected / at risk) | 50/157 | 56/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cardioplegia (N=157) | Microplegia (N=157)
Postoperative Acute Kidney Injury (Renal and urinary disorders) | 11 | 9 — Per STS Definition
Postoperative Hemodialysis (Renal and urinary disorders) | 10 | 8
Prolonged Ventilation (Respiratory, thoracic and mediastinal disorders) | 20 | 14 — STS Definition
Tracheostomy (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Reintervention due to MI (Cardiac disorders) | 0 | 1
Stroke (Nervous system disorders) | 4 | 2
Postoperative ECMO (Cardiac disorders) | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cardioplegia (N=157) | Microplegia (N=157)
Pneumonia (Infections and infestations) | 10 | 5 — STS Definition
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Postoperative Atrial Fibrillation (Cardiac disorders) | 38 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT05076604/Prot_SAP_000.pdf